CLINICAL TRIAL: NCT05739474
Title: Randomized, Double-blind, Comparative, Controlled Trial of Tolerability, Safety and Immunogenicity of the Flu-M Tetra Vaccine in Children Between 6 Months and 17 Years Old
Brief Title: Tolerability, Safety and Immunogenicity Trial of the Flu-M Tetra Vaccine in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FLМ-ТЕ-05-2021
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Influenza; Influenza, Human; Influenza Viral Infections; Vaccine Reaction
Keywords: Influenza; Flu; Vaccine; Vaccination; SPbSRIVS; Flu-M Tetra
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Flu-M Tetra vaccine, children aged 10 to 17 years old (Experimental): Сhildren will be vaccinated a single 0.5 mL dose of the Flu-M Tetra vaccine intramuscularly
  Interventions: Biological: Influenza vaccine [inactivated]
- VaxigripTetra vaccine, children aged 10 to 17 years old (Active Comparator): Сhildren will be vaccinated a single 0.5 mL dose of the VaxigripTetra vaccine intramuscularly
  Interventions: Biological: Influenza vaccine [inactivated]
- Flu-M Tetra vaccine, children aged 3 to 9 years old (Experimental): Сhildren will be vaccinated a single 0.5 mL dose of the Flu-M Tetra vaccine intramuscularly or double dose for volunteers who have not been vaccinated before
  Interventions: Biological: Influenza vaccine [inactivated]
- VaxigripTetra vaccine, children aged 3 to 9 years old (Active Comparator): Сhildren will be vaccinated a single 0.5 mL dose of the VaxigripTetra vaccine intramuscularly or double dose for volunteers who have not been vaccinated before
  Interventions: Biological: Influenza vaccine [inactivated]
- Flu-M Tetra vaccine, children aged 6 to 35 months old (Experimental): Сhildren will be vaccinated twice 0.25 mL dose of the Flu-M Tetra vaccine intramuscularly
  Interventions: Biological: Influenza vaccine [inactivated]
- VaxigripTetra vaccine, children aged 6 to 35 months old (Active Comparator): Сhildren will be vaccinated twice 0.25 mL dose of the VaxigripTetra vaccine intramuscularly
  Interventions: Biological: Influenza vaccine [inactivated]

INTERVENTIONS:
Biological: Influenza vaccine [inactivated] — solution for intramuscular injection, 1 dose (0.5 mL)
  Other Names: Flu-M Tetra Inactivated Split Quadrivalent Influenza Vaccine
  Arms: Flu-M Tetra vaccine, children aged 10 to 17 years old; Flu-M Tetra vaccine, children aged 3 to 9 years old; Flu-M Tetra vaccine, children aged 6 to 35 months old
Biological: Influenza vaccine [inactivated] — suspension for intramuscular and subcutaneous injection, 1 dose (0.5 mL)
  Other Names: VaxigripTetra (inactivated split influenza vaccine)
  Arms: VaxigripTetra vaccine, children aged 10 to 17 years old; VaxigripTetra vaccine, children aged 3 to 9 years old; VaxigripTetra vaccine, children aged 6 to 35 months old

SUMMARY:
The goal of this clinical trial is to assess tolerability, reactogenicity, safety and immunogenicity of the Flu-M Tetra vaccine as compared to the VaxigripTetra vaccine in terms of prevention of influenza in children aged 6 months to 17 years old inclusive.

DETAILED DESCRIPTION:
The trial will be conducted in three stages.

• Stage I Participants - children aged 10 to 17 years (10 years 0 months 0 days - 17 years 11 months 30 days), will be vaccinated a single 0.5 mL dose of the Flu-M Tetra vaccine or the VaxigripTetra vaccine intramuscularly.

Once reviewed by the Sponsor, the report will be submitted to the supervisory executive authorities alongside the notice of commencement of Stage II trial.

• Stage II Participants - children aged 3 to 9 years (3 years 0 months 0 days - 9 years 11 months 30 days), will be vaccinated a single 0.5 mL dose of the Flu-M Tetra vaccine or the VaxigripTetra vaccine intramuscularly (double dose for volunteers who have not been vaccinated before).

Once reviewed by the Sponsor, the report will be submitted to the supervisory executive authorities alongside the notice of commencement of Stage III trial.

• Stage III Participants - children aged 6 to 35 months (6 months 0 days - 35 months 30 days), will be vaccinated twice 0.25 mL dose of the Flu-M Tetra vaccine or the VaxigripTetra vaccine intramuscularly.

ELIGIBILITY:
Inclusion Criteria:

For volunteers aged 10 to 17 years:

* Healthy children of both sexes aged 10 to 17 years (10 years 0 months 0 days - 17 years 11 months 30 days);
* The availability of written and dated informed consent of the volunteer (children aged 14 to 17 years) and their parent / legally acceptable representative for participation in the trial;
* If the volunteer has sexual relations, effective contraception methods must be used during the 30 days preceding vaccination and consent must be obtained to continue using these contraceptive methods during the trial and for two months after vaccination;
* The girls with menses in the medical history shall have a negative pregnancy test result.

For volunteers aged 3 to 9 years:

* Healthy children of both sexes aged 3 to 9 years (3 years 0 months 0 days - 9 years 11 months 30 days);
* The availability of written and dated informed consent of a parent / legally acceptable representative for participation in the trial;

For volunteers aged 6 to 35 months:

* Healthy children of both genders aged 6 to 35 months, inclusive (6 months 0 days - 35 months 30 days);
* The availability of written and dated informed consent of a parent / legally acceptable representative for participation in the trial.
* The trial subject of the was born full-term, with the Apgar score of 7-10 points.

For all volunteers:

The ability of a volunteer's parents / legally acceptable representatives to perform the requirements of the Protocol (i.e., fill out the Patient Diary, attend visits together with the volunteer).

Exclusion Criteria:

1. History of influenza (including in mothers for children aged 6 to 35 months) or previous influenza vaccination during 6 months before the trial;
2. Vaccination of the pregnant woman in the 2nd-3rd trimester (for the age group of 6 - 35 months) with an influenza vaccine
3. Positive result of the SARS-CoV-2 test;
4. Vaccination with any vaccine less than 30 days before participating in the trial or scheduled vaccination with any vaccine within 30 days after vaccination with the trial vaccines;
5. A serious post-vaccination reaction (temperature above 40 °C, hyperemia or edema more than 8 cm in diameter at the injection site) or complications (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions accompanied or not accompanied by a fever due to any previous vaccination), encephalopathy;
6. Allergic reactions to vaccine components or any previous vaccination;
7. History of allergic reaction to chicken protein;
8. History of cancer, leukemia, tuberculosis, autoimmune diseases;
9. Carriage of HIV, syphilis, hepatitis B and C in the medical history, including by parents / legally acceptable representatives;
10. Children who received immunoglobulin products or transfusions of whole blood or its components less than 3 months before the start of the trial;
11. Long-term use (more than 14 days) of any immunomodulating medicines less than 3 months before the start of the trial;
12. Any confirmed or suspected immunosuppressive or immunodeficiency condition;
13. History of chronic diseases of the cardiovascular, bronchopulmonary, endocrine systems, blood in the acute stage (recovery less than 4 weeks before vaccination) or in the decompensation stage;
14. Children with hemophilia who may develop bleeding after intramuscular injection;
15. History of progressive neurological pathology, convulsive syndrome, afebrile convulsions;
16. History of acute infectious diseases (fever ≥ 37.5°С): recovery less than 2 weeks before vaccination;
17. Participation in another clinical trial less than 3 months before the start of the trial;
18. History of mental illness of the child and the volunteer's parents;
19. The history of the volunteer's parent / legally acceptable representative being registered with a tuberculosis dispensary and/or a narcological dispensary;
20. Maternal history of drug use or alcohol abuse during pregnancy and/or breastfeeding;
21. Pronounced congenital malformations in a child;
22. Suspected developmental delay in a child.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 948 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Geometric mean titer (GMT) ratio of antibodies for each virus strain (A (H1N1), A (H3N2) and B) | Baseline (day 1) and 28 days after vaccination (Stage I, II, III) and revaccination (Stage II, III)
  Geometric mean titer (GMT) of antibodies in the blood serums of vaccinated participants in haemagglutination inhibition assay

SECONDARY OUTCOMES:
Change from Baseline Seroconversion factor for each virus strain (A (H1N1), A (H3N2) and B) | Baseline (day 1) and 28 days after vaccination (Stage I, II, III) and revaccination (Stage II, III)
  Seroconversion factor is an increase in the geometric mean titers of antibodies at Day 28 vs. the baseline level, expressed in the fold rise
Change from Baseline Seroprotection rate for each virus strain (A (H1N1), A (H3N2) and B) | Baseline (day 1) and 28 days after vaccination (Stage I, II, III) and revaccination (Stage II, III)
  Seroprotection rate refers to the percentage of subjects with a generated protective HA titer (at least 1:40) vs. the baseline level
Change from Baseline Seroconversion rate for each virus strain (A (H1N1), A (H3N2) and B) | Baseline (day 1) and 28 days after vaccination (Stage I, II, III) and revaccination (Stage II, III)
  Seroconversion rate refers to the percentage of subjects who have a prevaccination titer of influenza haemagglutinin antibody titer (HA titer) ≤ 1:10 and a post-vaccination HA titer ≥ 1:40 or a prevaccination HA titer > 1:10 and at least a 4-fold increase in post-vaccination HA titer vs. the baseline
Incidence of immediate adverse events (allergic reactions) | 2 hours after vaccination
Incidence of local adverse events | 7 days after vaccination
Incidence of systemic adverse events | 7 days after vaccination
Incidence of other adverse reactions | Days 8 to 28 after vaccination
Incidence of severe adverse events | Days 1 to 28+3 (for participants with 1 vaccination), Day 1 to 56±3 (for participants with vaccination and revaccination)
Withdrawal of a volunteer from the trial due to development of an AE/SAE associated with the use of the trial products | Days 1 to 28+3 (for participants with 1 vaccination), Day 1 to 56±3 (for participants with vaccination and revaccination)
Number of participants with abnormal physical examination findings | Days 1, 3, 7, 28+3 (for participants with 1 vaccination), Days 1,3,7,28+3,56±3 (for participants with vaccination and revaccination)
  Physical examination of volunteers includes an interview, discovery of complaints and symptoms, when required, palpation, auscultation, percussion.
  It is necessary to conduct an examination of the following organs and systems: skin, mucosa, eyes, oral cavity and pharynx, lungs/chest, heart/cardiovascular system, abdominal organs, nervous system, lymph nodes, musculoskeletal system
Number of participants with abnormal changes in vital signs - Blood pressure (BP) | Days 1, 3, 7, 28+3 (for participants with 1 vaccination), Days 1,3,7,28+3,56±3 (for participants with vaccination and revaccination)
  BP is assessed in children aged 36 months and older. BP measurements include the systolic and diastolic blood pressure.
Number of participants with abnormal changes in vital signs - Heart rate (HR) | Days 1, 3, 7, 28+3 (for participants with 1 vaccination), Days 1,3,7,28+3,56±3 (for participants with vaccination and revaccination)
  HR is measured using a phonendoscope at the apex of the heart during 1 minute.
Number of participants with abnormal changes in vital signs - Respiratory rate (RR) | Days 1, 3, 7, 28+3 (for participants with 1 vaccination), Days 1,3,7,28+3,56±3 (for participants with vaccination and revaccination)
  RR is counted with a hand placed on the child's chest or abdomen or by holding a stethoscope at the child's nose. The measurement is conducted during one minute.
Number of participants with abnormal changes in vital signs - Body temperature | Days 1, 3, 7, 28+3 (for participants with 1 vaccination), Days 1,3,7,28+3,56±3 (for participants with vaccination and revaccination)
  The body temperature is measured with a digital thermometer.
Number of participants with clinically significant abnormalities - Complete blood count (CBC) | Days 1, 3
  Hemoglobin, Hematocrit, Erythrocytes, Leukocytes, Leukocytic Formula, Platelets, Erythrocyte Sedimentation Rate (ESR)
Number of participants with clinically significant abnormalities - Biochemical blood test (BBT) | Days 1, 3
  ALT, AST, Alkaline Phosphatase, Total Bilirubin, Total Protein, Urea, Glucose
Number of participants with clinically significant abnormalities - Urinalysis | Days 1, 3
  pH, Color, Relative Density/Specific Gravity, Protein, Glucose, Red Blood Cells, White Blood Cells
Number of participants with abnormal changes of total IgE | Days 1, 3
Number of participants with abnormal neurological examinations | Days 1, 3, 7, 28+3 (for participants with 1 vaccination), Days 1,3,7,28+3,56±3 (for participants with vaccination and revaccination)

CONTACTS AND LOCATIONS:
Overall Officials: Ellina Ruzanova, PhD, Study Director — St. Petersburg Research Institute of Vaccines and Sera
Locations (7):
- Russia (7):
  - State Autonomous Health Care Institution "Engels City Clinical Hospital No1", Engel's
  - Llc "Olla-Med", Moscow
  - LLC "Professorskaya Clinica", Perm
  - State Budgetary Healthcare Institution of the Perm Territory "City Children's Clinical Clinic No. 5", Perm
  - LLC PiterClinica, Saint Petersburg
  - LLC "DNA Research Center", Saratov
  - State Autonomous Health Care Institution of the Sverdlovsk Region "Children's City Clinical Hospital No. 11", Yekaterinburg